CLINICAL TRIAL: NCT02163707
Title: Pharmacokinetics of Psilocybin in Normal Adult Volunteers
Brief Title: UW Psilocybin Pharmacokinetics Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0998; A561000 (Other: UW Madison); PHARM\PHARMACY\PHARMACY (Other: UW Madison)
Record Dates: First submitted 2014-06-03; First posted 2014-06-16 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Healthy
Keywords: Psilocybin; Pharmacokinetics
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Psilocybin Dose 1 (Other): 0.3 mg/kg (approximately 20mg/70kg)
  Interventions: Drug: Psilocybin
- Psilocybin Dose 2 (Other): 0.45 mg/kg (approximately 30 mg/70 kg)
  Interventions: Drug: Psilocybin
- Psilocybin Dose 3 (Other): 0.6 mg/kg (approximately 40 mg/70 kg)
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Dose 1: 0.3 mg/kg (approximately 20mg/70kg) Dose 2: 0.45 mg/kg (approximately 30 mg/70 kg) Dose 3: 0.6 mg/kg (approximately 40 mg/70 kg)

SUMMARY:
Psilocybin is a naturally occurring psychedelic compound produced by more than 200 species of mushrooms, collectively known as psilocybin mushrooms. Psilocybin (4-phosphoroyloxy-N,N-dimethyltryptamine) is a hallucinogenic tryptamine that was first isolated from Psilocybe mushrooms in 1957. The objective of this Phase I clinical trial is to determine the pharmacokinetics of oral doses of psilocybin in normal, healthy adults. The study is performed in support of Phase II and Phase III studies of psilocybin for the treatment of refractory anxiety associated with incurable cancer, as well as other possible indications. Psilocybin is at present not an FDA-approved drug.

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to determine the pharmacokinetics of an extemporaneous oral formulation of psilocybin in normal, healthy adults. This study is intended to add to the existing body of modern clinical research on psilocybin to support future multi-institutional Phase III clinical trials seeking to decrease anxiety and depression in patients with incurable cancer. The long-term goal of this research is to submit a successful new drug application for psilocybin to the FDA.

Subjects will initially take one 0.3 mg/kg (approximately 20mg/70kg) oral dose of psilocybin to initiate an eight hour chaperoned outpatient experience. After eight hours of outpatient sampling, the subject will be transported across the street to the UW Institute for Clinical and Translational Research Clinical Research Unit (ICTR CRU) for an overnight stay and additional blood and urine sampling. Pre- and post-treatment psychologic preparation and debriefing interviews will be required.

A minimum of four weeks after the first dose, the subject will receive a second oral dose of psilocybin at the higher dose of 0.45 mg/kg (approximately 30 mg/70 kg). This dosing will again take place in an attended, structured setting with timed blood and urine samples obtained both in the School of Pharmacy (0-8 hours) and in the UW Clinical Research Unit (8-24 hours). A minimum of four weeks after the second dose, the subject will receive a third oral dose of psilocybin at the highest dose of 0.6 mg/kg (approximately 40 mg/70 kg). This dose will again take place in an attended, structured setting with timed blood and urine samples obtained both in the School of Pharmacy (0-8 hours) and in the UW Clinical Research Unit (8-24 hours).

12-lead ECGs will be obtained at specified time points before and during each treatment period. Throughout the duration of drug action for each dose participants will be attended by two trained monitors, and a physician will available during the entire 24 hour treatment and sampling period.

Subjects who have been administered the first dose but decline to receive any subsequent doses will remain evaluable. At that time their active study participation will end.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 - 80 years
* Able to read, speak, and understand spoken English
* Self-report of at least one prior positive hallucinogen drug experience that included a meaningful altered state of consciousness. Hallucinogenic substances can include psilocybin, LSD, or other classic hallucinogens.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 based upon CRU NP or study physician physical exam, which indicates a subject is fully functioning.
* A woman of childbearing potential must agree to practice an effective means of birth control during their participation in the clinical trial, up to and including the 90 day follow-up after their last psilocybin dose. Birth control method and written agreement to practice this method throughout the duration of the study will be documented on the Medical History Case Report Form. Effective contraception is defined as the regular use of one of the following:

  * Established use of oral, injected, or implanted hormonal methods of contraception
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  * Barrier methods: Condom or Occlusive cap used with a spermicide
  * female sterilization/hysterectomy (with documentation of surgery)
  * post-menopausal (>12 months since last menses at the time of screening)
  * Male sterilization (with post-vasectomy documentation)
  * True abstinence
* Ability and willingness to adhere to study requirements, including attending all study visits, preparatory and follow-up sessions, and completing all study evaluations.
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages and tobacco, within 24 hours of each drug administration. The exception is caffeine.
* Participants will be required to be non-smokers.

Exclusion Criteria:

* Estimated creatinine clearance <30 ml/min, using the Cockcroft Gault equation and actual body weight.
* Clinically significant abnormal chemistry or hematologic laboratory results (from a screen of Complete Blood Count with Differential and Comprehensive Metabolic Panel), using the UWHC core lab reference intervals.
* Females of childbearing potential with positive urine pregnancy at screening or the day of the first treatment.
* Clinically significant abnormalities in physical examination.
* Inadequately treated hypertension (systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg).
* Personal history of primary psychotic disorder (unless substance-induced or due to a medical condition), bipolar affective disorder Type I or Type II, or schizophrenia.
* First or second-degree family history of primary psychotic disorder, bipolar affective disorder Type I, bipolar affective disorder Type II, or schizophrenia.
* Substance abuse or dependency within the past five years.
* Suicidal ideation or attempt within the past 30 days and/or any prior suicidal ideation/attempt that the study physician and PI feel makes the participant unsuitable for the study.
* Urine drug test containing non-prescribed drugs of abuse (non-prescribed opioids, benzodiazepines, amphetamines, phencyclidine, cocaine) at screening and day of first treatment. Urine cannabinoid concentrations >50 ng/ml will suggest heavy marijuana use, and will be a threshold for excluding potential subjects.
* Current use of monoamine oxidase inhibitors or dopaminergic antagonists. Any prohibited agents must have been stopped at least 5x the elimination half-life of the specific drug.
* Subject does not have a local support person that is available during their 24 hour treatment and observation period.
* Concurrent or recent (within 5 years) history of major depression, obsessive-compulsive disorder, panic disorder, anorexia nervosa, or bulimia nervosa.
* Poor venous access.
* Known acute coronary syndrome or angina.
* Evidence of ischemic disease or ventricular arrhythmias on screening ECG.
* Cardiac conduction defects on screening ECG.
* Cardiac transplantation as determined by self-report during review of medical history.
* Lactose intolerance (excipient in psilocybin capsules)
* Type I or insulin-dependent Type II diabetes.
* Prescription medicine requiring dosing during the 8 hours of drug action.
* Current or recent (past 5 years) seizure disorder as determined by self-report during medical history and physical exam.
* Chronic or frequent migraines.
* Regular or frequent use of benzodiazepines.
* Attention Deficit Hyperactivity Disorder (ADHD) or Attention Deficit Disorder (ADD).
* Regular or frequent use of stimulants.
* Generalized Anxiety Disorder (GAD).
* Post-Traumatic Stress Disorder (PTSD).
* Neuroleptic medications.
* Any physical or psychological symptom, based on the clinical judgment of the study physician and/or psychologist , that would make a participant unsuitable for the study.
* Any use of a medication(s), based on the clinical judgment of the study physician, that would make a participant unsuitable for the study.
* Any finding(s), based on the screening process, that the PI feels makes the participant unsuitable for the study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Determine the concentrations of psilocin following escalating doses of psilocybin | 12 months
  Determine the AUC of psilocin in plasma following single doses of 0.3, 0.45, and 0.6 mg/lg psilocybin, the precursor to psilocin.

SECONDARY OUTCOMES:
Characterize any non-linearity in the pharmacokinetics of psilocybin and psilocin. | 12 months
  Quantitate any non-linearity of the plasma AUC of psilocybin and its active metabolite psilocin after escalation doses of psilocybin.
Determine the effect of kidney function on psilocin pharmacokinetics. | 12 months
  Use urine and plasma collections to quantitate the relative renal clearance of creatinine and psilocin to characterize the dependency of renal clearance of psilocin upon the glomerular filtration rate. Variation in renal function will arise from the range of ages in subjects; subjects are not selected or grouped based upon renal function.
Characterize the incidence and severity of adverse events associated with escalating doses of psilocybin in normal adults. | 12 months
  The incidence and severity of expected and unexpected adverse events will be collected using the NCI Common Toxicity Criteria for Adverse Events (CTCAE) v4 during and in treatment follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hutson, PharmD, Principal Investigator — University of Wisconsin, School of Pharmacy
Locations (1):
- University of Wisconsin, School of Pharmacy, Madison, Wisconsin, United States

REFERENCES:
- [Result] Brown RT, Nicholas CR, Cozzi NV, Gassman MC, Cooper KM, Muller D, Thomas CD, Hetzel SJ, Henriquez KM, Ribaudo AS, Hutson PR. Pharmacokinetics of Escalating Doses of Oral Psilocybin in Healthy Adults. Clin Pharmacokinet. 2017 Dec;56(12):1543-1554. doi: 10.1007/s40262-017-0540-6. PMID 28353056
- [Result] Nicholas CR, Henriquez KM, Gassman MC, Cooper KM, Muller D, Hetzel S, Brown RT, Cozzi NV, Thomas C, Hutson PR. High dose psilocybin is associated with positive subjective effects in healthy volunteers. J Psychopharmacol. 2018 Jul;32(7):770-778. doi: 10.1177/0269881118780713. Epub 2018 Jun 27. PMID 29945469